CLINICAL TRIAL: NCT01754298
Title: Retro Versus Trans Articular Drilling for Juvenile Osteochondritis Dissecans of the Knee: A Multicenter, Randomized Controlled Trial
Brief Title: Study of Two Surgical Drilling Techniques to Treat Juvenile Osteochondritis Dissecans of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Pediatric Orthopaedic Society of North America (Other); University of Pennsylvania (Other); Tennessee Orthopedic Alliance (Other); Children's Hospital Medical Center, Cincinnati (Other); Children's Hospital and Health System Foundation, Wisconsin (Other); Washington University School of Medicine (Other); The Hospital for Sick Children (Other); Children's Hospital of Philadelphia (Other); Kaiser Permanente (Other); Rady Children's Hospital, San Diego (Other); St. Luke's Children's Hospital (Other); Medical College of Wisconsin (Other); Connecticut Children's Medical Center (Other); Hospital for Special Surgery, New York (Other)
Responsible Party: Principal Investigator, Benton Heyworth, Instructor in Orthopaedic Surgery, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-P00004016
Record Dates: First submitted 2012-12-16; First posted 2012-12-21 (Estimated); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Juvenile Osteochondritis Dissecans
Keywords: osteochondritis dissecans (OCD); juvenile osteochondritis dissecans (JOCD); knee osteochondritis dissecans; retro-articular drilling; trans-articular drilling; stable osteochondritis dissecans lesion
MeSH Terms: conditions — Osteochondritis Dissecans

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Retro-articular drilling (Active Comparator): Retro-articular drilling goes through the cortical margin of the affected condyle, thereby sparing the articular surface and physes.
  Interventions: Procedure: Retro-articular drilling
- Trans-articular drilling (Active Comparator): Trans-articular drilling penetrates the articular cartilage through multiple sites to create subchondral penetrations.
  Interventions: Procedure: Trans-articular drilling

INTERVENTIONS:
Procedure: Retro-articular drilling — * Drilling must be performed under AP and lateral fluoroscopic guidance, with no additional drilling in 'trans-articular', or intra-articular trans-condylar fashion.
  * Use a 0.045 K-wire for drilling.
  * Minimum of 8 wire passes per square centimeter with no maximum number of wire passes.
  Other Names: antero-grade; extra-articular
  Arms: Retro-articular drilling
Procedure: Trans-articular drilling — * Drilling must be performed, under arthroscopic visualization, directly through the articular cartilage, with no additional drilling in 'retro-articular', 'extra-articular', or trans-condylar (through the intercondylar notch)
  * Use a 0.045 K-wire for drilling
  * A minimum 4 wire passes per square centimeter, with a maximum of 5 wire passes per square centimeter
  Other Names: antero-grade; extra-articular
  Arms: Trans-articular drilling

SUMMARY:
The purpose of this study is to compare the functional, clinical and radiographic outcomes associated with trans-articular drilling versus retro-articular drilling, two commonly employed techniques of operative treatment for stable forms of juvenile osteochondritis dissecans (JOCD) lesions. This study also aims to better define the natural history of this condition in its most commonly identified pathological state (as a stable lesion) following surgical intervention by determining the rate of radiographic healing and any need for secondary surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of JOCD,
* Lesion located on the lateral aspect of the medial femoral condyle,
* Lesion considered stable based on MRI,
* Patient deemed skeletally immature based on MRI,
* Completed a course of conservative therapy.

Exclusion Criteria:

* Significant concomitant knee pathology (AVN, fracture, inflammatory arthritis, ACL tear, discoid/meniscal tear, etc.)
* Lesion healed sufficiently and surgery is not recommended,
* Prior surgery on the affected knee,
* Diagnosis of metabolic bone disorder (e.g. osteogenesis imperfecta),
* Diagnosis of sickle cell disease,
* History of prolonged corticosteroid or chemotherapy treatment,

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 91 (Actual)
Dates: Start 2013-01-18 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Physical functioning measured by the Pedi-IKDC (International Knee Documentation Committee) total score | One year post-surgery

SECONDARY OUTCOMES:
Activity level as measured by the Marx Activity Scale | One year post-surgery
Physical functioning as measured by the Pedi-IKDC total score | Two years post-surgery
Time to lesion healing | 3 months to 2 years post-surgery
  Lesion healing will be assessed by x-ray at multiple time points

OTHER OUTCOMES:
Surgical complications | 1 week to 1 year post-surgery
  Inadvertent displacement of OCD fragment; damage to articular cartilage and physes

CONTACTS AND LOCATIONS:
Overall Officials: Benton Heyworth, M.D., Principal Investigator — Boston Children's Hospital
Locations (14):
- United States (13):
  - Kaiser Permanente Los Angeles, Los Angeles, California
  - Rady Children's Hospital, San Diego, California
  - Rocky Mountain Hospital for Children, Centennial, Colorado
  - Connecticut Children's Medical Center, Farmington, Connecticut
  - St. Luke's Children's Hospital, Boise, Idaho
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Hospital for Special Surgery, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Tennessee Orthopaedic Alliance, Nashville, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Heyworth BE, Ganley TJ, Liotta ES, Hergott KA, Miller PE, Wall EJ, Myer GD, Nissen CW, Edmonds EW, Lyon RM, Chambers HG, Milewski MD, Green DW, Weiss JM, Wright RW, Polousky JD, Nepple JJ, Carey JL, Kocher MS; ROCK Group; Shea KG. Transarticular Versus Retroarticular Drilling of Stable Osteochondritis Dissecans of the Knee: A Prospective Multicenter Randomized Controlled Trial by the ROCK Group. Am J Sports Med. 2023 May;51(6):1392-1402. doi: 10.1177/03635465231165290. Epub 2023 Apr 11. PMID 37039536
- See also: Research in OsteoChondritis of the Knee, OCD Study Group of North America — https://kneeocd.org//